CLINICAL TRIAL: NCT03550573
Title: 3D Non-invasive Myocardial Electrical Propagation Mapping as a New Tool to Predict Sudden Death Risk in Patients With Hypertrophic Cardiomyopathy: A Pilot Study
Brief Title: 3D Non-invasive Myocardial Electrical Propagation Mapping as a New Tool to Predict Sudden Death Risk in Patients With Hypertrophic Cardiomyopathy
Acronym: 3D-CMH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL17_0657; ID-RCB (Other: 2018-A00211-54)
Record Dates: First submitted 2018-05-25; First posted 2018-06-08 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Hypertrophic cardiomyopathy; sudden death; 3D mapping
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Death, Sudden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hypertrophic cardiomyopathy without sudden death history (Experimental)
  Interventions: Device: CardioInsight™ Noninvasive 3D Mapping System
- hypertrophic cardiomyopathy with sudden death history (Experimental)
  Interventions: Device: CardioInsight™ Noninvasive 3D Mapping System

INTERVENTIONS:
Device: CardioInsight™ Noninvasive 3D Mapping System — The CardioInsight system uses a proprietary, single-use, disposable multi-electrode vest to capture electrical signals from the body surface. The CardioInsight software provides various cardiac signal analyses and displays interactive 3-D color maps including activation, voltage, composite and phase maps. The vest wearing is coupled with a CT scan.
  This exam will be performed only at baseline visit.

SUMMARY:
Hypertrophic cardiomyopathy (HCM) is very common. The thickened heart muscle can disrupt the normal functioning of the heart's electrical system, resulting in fast or irregular heartbeats. Today, there are no reliable means to identify HCM patients at risk of sudden death. The CardioInsight™ has recently been developed by Medtronic for non-invasive advanced cardiac mapping system. The CardioInsight™ Noninvasive 3D Mapping System is a non-invasive mapping system that collects chest ECG signals and combines these signals with CT scan data to produce and display simultaneous, bi-atrial and biventricular, 3-D cardiac maps.

It is a monocentric, prospective, comparative and analytical study. 20 HCM patients will be recruited in the National Reference Center for inherited cardiac diseases of Lyon. The 3D-propagation maps of 10 well phenotyped and genotyped HCM patients with previous VF (ventricular fibrillation) will be compared to 10 HCM patients without previous VF.

After consent signed, Holter ECG, scanner and CardioInsightTM 3D_ECG mapping will be planned in the month following the inclusion. 12-lead ECG, 24h holter ECG, cardiac scanner will be performed as standard procedure of each center in the current health care of the patient.

The widespread screening of HCM patients with 3D high-density noninvasive mapping should improve the risk-benefit ratio of implantable defibrillator therapy. It is expected that more patients at risk will benefit from this device.

ELIGIBILITY:
Inclusion criteria :

* HCM patient confirmed by echocardiogram.
* Patient who signed the consent.
* Patient benefiting from a social insurance system or a similar system

Exclusion Criteria:

* pregnant women,
* left ventricular dilation (diastolic >60 mm diameter) and/or left ventricular systolic dysfunction (LVEF <55%),
* prior cardiac surgery,
* atrial fibrillation,
* renal disease (serum creatinine >2.0 mg/dl),
* primary cardiac valve disease
* coronary artery disease
* Previous recent cardiac scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-09-23 (Actual)

PRIMARY OUTCOMES:
Identification of specific markers of risk of sudden death in HCM patients from the maps created by the combination of CT and signal data. | Month 1
  The CardioInsight system uses a proprietary, single-use, disposable multi-electrode vest to capture electrical signals from the body surface. The CardioInsight software provides various cardiac signal analyses and displays interactive 3-D color maps including activation, voltage, composite and phase maps. The use of the CardioInsight system is correlated with a CT scan.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Louis Pradel, Bron, France

IPD SHARING:
Plan to Share IPD: Undecided